CLINICAL TRIAL: NCT02481817
Title: Treatment Alternatives in Adult Rare Disease; Assessment of Options in Idiopathic Subglottic Stenosis North American Airway Collaborative PR-02 Study (NoAAC PR-02 Study)
Brief Title: Treatment Alternatives in iSGS (NoAAC PR-02 Study)
Acronym: NoAAC PR-02
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); The Cleveland Clinic (Other); University of Utah (Other); Johns Hopkins University (Other); Vanderbilt University (Other); University of Virginia (Other); Massachusetts Eye and Ear Infirmary (Other); Oregon Health and Science University (Other); University of Washington (Other); University of California, San Francisco (Other); University of California, Los Angeles (Other); University of California, San Diego (Other); University of Colorado, Denver (Other); Baylor College of Medicine (Other); Louisiana State University Health Sciences Center in New Orleans (Other); Charing Cross Hospital (Other); University of Alabama at Birmingham (Other); University of Wisconsin, Madison (Other); University of Michigan (Other); University of Nebraska (Other); University of Iowa (Other); University of Texas (Other); Duke University (Other); University of North Carolina (Other); Augusta University (Other); University of Sydney (Other); North American Airway Collaborative (Unknown); University of California, Irvine (Other); University of Pittsburgh (Other); Loma Linda University (Other); Stanford University (Other); University of Cincinnati (Other); Emory University (Other); Ohio State University (Other); University of Southern California (Other); Temple University (Other); Medical College of Wisconsin (Other); Landspitali University Hospital (Other); Bastian Voice Institute (Unknown); NYU Langone Health (Other); Mayo Clinic (Other); University of Miami (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Alexander Gelbard, MD, Assistant Professor, Department of Otolaryngology, Vanderbilt University Medical Center
Other Study IDs: 150917
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Subglottic Stenosis (iSGS)
MeSH Terms: conditions — Idiopathic subglottic tracheal stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens collected during routine standard of care from each patient (such as tracheal biopsies obtained during surgery, or surgical specimens generated thru open reconstructive surgeries), will be annotated in the EDC with such data including specimen collection, specimen type (e.g., frozen biopsy tissue; FFPE block), and storage location. We may examine excess tissue obtained at standard of care surgical biopsy. Additionally if blood is collected during standard of care (i.e., medically indicated labs, operative or office-based procedures), we will ask participants to provide a one-time, 30 mL blood specimen for research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iSGS patients: Participants will receive standard of care treatment at the respective center and will be followed longitudinally for symptom changes, need for further treatment, complications, and will have Patient-reported outcomes (PROs) administered at a priori determined intervals.
  Interventions: Procedure: Endoscopic dilation of subglottic stenosis; Procedure: Endoscopic resection of the stenosis; Procedure: Tracheal Resection

INTERVENTIONS:
Procedure: Endoscopic dilation of subglottic stenosis — This is accomplished with rigid instruments or inflatable balloons.
Procedure: Endoscopic resection of the stenosis — This is accomplished with C02 lasers and paired with prolonged medical therapy after surgery.
Procedure: Tracheal Resection — Resection of the affected tracheal segment with end-to-end anastomosis
  Other Names: Cricotracheal Resection; Open Airway Surgery

SUMMARY:
The study is aimed at answering the questions; (1) How well do the most commonly used treatments in iSGS work? and (2) What quality-of-life trade-offs are associated with each approach?

With the results of this trial, the investigators hope to provide information to iSGS patients: (1) Given my personal characteristics, conditions, and preferences, what should I expect will happen to me? and (2) What are my options, and what are the potential benefits and harms of these options?

DETAILED DESCRIPTION:
Idiopathic subglottic stenosis (iSGS) is a rare disease in which the trachea narrows for no known reason. Although uncommon (with an estimated incidence of 1:400,000 persons per year), both the disease and its therapies profoundly affect patients' ability to breathe, communicate and swallow. Breathing difficulties (i.e. dyspnea) is the hallmark symptom and the primary cause of death and disability. However, patients can also experience debilitating voice changes and swallowing problems due to the condition or its treatment.

People with this disease often require several surgeries per year. A variety of treatments have been advanced to manage iSGS but are generally categorized into: 1) endoscopic dilation of the tracheal stenosis (accomplished with rigid instruments or inflatable balloons); 2) endoscopic resection of the stenosis (with prolonged medical therapy after surgery); or 3) open neck surgery with resection of the affected tracheal segment with end-to-end anastomosis. Each patient can require repeated surgeries to keep their trachea open, which increases odds of treatment side effects and complications. All approaches have unique and often disabling associated side effects, which can significantly affect a patient's quality of life.

Because the disease is rare, it is difficult for patients to find good information so that they can understand the spectrum of treatment options. This is particularly difficult because most patients present with severe breathing trouble and need treatment quickly, limiting their ability to explore options. Additionally, there is a general lack of high-quality, reliable, and accessible data to inform individual patient decision-making. Imperfect information and limited evidence on treatment outcomes complicate patient decision-making as they try to balance survival, symptoms, and quality of life considerations.

Beyond the gaps in understanding the relative effectiveness of the different treatments available, no studies have explored functional outcomes in iSGS (i.e. how well patients breathe, speak, and swallow after treatments). These endpoints are important to patients and are arguably a primary determinant in decision-making. Direct engagement with patients is critical to understand these quality of life considerations, since patient and physician perspectives aren't always the same. For example, results show that endoscopic dilation is associated with a higher rate of disease recurrence and thus need for repeated surgery. Meanwhile, open tracheal resection is a major surgery with significant immediate perioperative risks and has been associated with alterations in voice and swallowing. Open tracheal resection appears to reduce the risk of disease recurrence, but the degree of benefit, and the trade-offs associated with this approach are unanswered questions.

The proposed study from the North American Airway Collaborative (NoAAC PR- 02) is designed to fill this void. Our prospective study will directly compare the effectiveness of standard of care treatments and assess their associated quality of life tradeoffs in iSGS patients.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age.
* The lesion must involve the subglottis.

Exclusion Criteria:

* Less than 18 years of age
* Patients without capacity to consent for themselves
* History of significant laryngotracheal traumatic injury.
* History of endotracheal intubation or tracheotomy within 2 years of presentation.
* Major anterior neck surgery.
* History of neck irradiation.
* History of caustic or thermal injuries to the laryngotracheal complex.
* History of a clinically diagnosed vasculitis or collage vascular disease.
* Positive antinuclear cytoplasmic antibody titers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All clinically confirmed iSGS patients at the participating institutions are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1239 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Treatment Effectiveness: Time to recurrent procedure | 3 years
Treatment Effectiveness: Need for tracheostomy | 3 years

SECONDARY OUTCOMES:
QOL | 3 years
  Patient quality of life assessment: voice (VHI-10)
QOL | 3 years
  Patient quality of life assessment: dysphagia (EAT-10)
QOL | 3 years
  Patient quality of life assessment: breathing (COPD dyspnea)
QOL | 3 years
  Patient quality of life assessment: general quality of life (SF-12)
Patient Reported Outcome | 3 years
  Non-traditional PRO focused on social support
Patient Reported Outcome | 3 years
  Non-traditional PRO focused on fear of disease recurrence
Patient Reported Outcome | 3 years
  Non-traditional PRO focused on disease anxiety and burden
Patient Reported Outcome | 3 years
  Non-traditional PRO focused on participatory decision-making style

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Gelbard, MD, Principal Investigator — Vanderbilt University Medical Center; David O. Francis, MD, MS, Study Chair — Vanderbilt University Medical Center
Locations (42):
- United States (39):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - University of California Irvine, Irvine, California
  - Loma Linda University Health Care, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Bastian Voice Institute, Downers Grove, Illinois
  - University of Iowa, Iowa City, Iowa
  - Louisiana State University, Baton Rouge, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - Harvard Medical School -Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - New York University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Cincinatti, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University of Sydney, St Leonards, Australia
- Landspitali University Hospital, Reykjavik, Iceland
- Charing Cross Hospital, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gelbard A, Shyr Y, Berry L, Hillel AT, Ekbom DC, Edell ES, Kasperbauer JL, Lott DG, Donovan DT, Garrett CG, Sandhu G, Daniero JJ, Netterville JL, Schindler JS, Smith ME, Bryson PC, Lorenz RR, Francis DO. Treatment options in idiopathic subglottic stenosis: protocol for a prospective international multicentre pragmatic trial. BMJ Open. 2018 Apr 10;8(4):e022243. doi: 10.1136/bmjopen-2018-022243. PMID 29643170

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT02481817/Prot_SAP_000.pdf